CLINICAL TRIAL: NCT01233154
Title: Effect of a L. Paracasei Strain on Grass Pollen Allergic Rhinitis Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07.27.NRC
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L. paracasei (Experimental): L. paracasei
  Interventions: Dietary Supplement: probiotic
- L. acidophilus + B. lactis (Experimental): L. acidophilus + B. lactis
  Interventions: Dietary Supplement: probiotic

INTERVENTIONS:
Dietary Supplement: probiotic
  Arms: L. paracasei
Dietary Supplement: probiotic
  Arms: L. acidophilus + B. lactis

SUMMARY:
Various studies in animal and humans have shown a potential beneficial effect of probiotics consumption on allergy. However few studies exist that document their efficacy for upper airways allergies such as allergic rhinitis. The objective of this study is to investigate the effect of short-term oral administration of a L. paracasei or of a blend of 2 probiotics (L. acidophilus + B. lactis) on a nasal provocation test (NPT) with grass pollen, performed out of the pollen season. Adult volunteers with allergic rhinitis are enrolled in a randomized, double-blind study, based on two 4-weeks cross-over periods of product consumption separated by a washout period of 6-8 weeks. Objective and subjective clinical parameters of NPT as well as systemic and nasal immunological markers are compared before and after each treatment.

ELIGIBILITY:
Inclusion Criteria:

* age 18-40 years old
* history of allergic rhinitis during the latest grass pollen season confirmed by a positive skin prick test to grass pollen (wheal diameter > 3mm) and a positive response to a NPT with grass pollen (combined nasal reaction threshold <= 10000 standardized quality units/ml at the screening phase

Exclusion Criteria:

* any medical condition that could influence the study (pregnancy, viral or bacterial airway infection, active allergic rhinitis)
* uncontrolled asthma (peak expiratory flow <20% of volunteer's best personal value)
* treatment with antihistamine or antibiotic treatment less than two weeks before enrolment or during the trial

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-10; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Nasal reaction threshold when provocation test with allergens | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

REFERENCES:
- [Result] Perrin Y, Nutten S, Audran R, Berger B, Bibiloni R, Wassenberg J, Barbier N, Aubert V, Moulin J, Singh A, Magliola C, Mercenier A, Spertini F. Comparison of two oral probiotic preparations in a randomized crossover trial highlights a potentially beneficial effect of Lactobacillus paracasei NCC2461 in patients with allergic rhinitis. Clin Transl Allergy. 2014 Jan 6;4(1):1. doi: 10.1186/2045-7022-4-1. PMID 24393277